CLINICAL TRIAL: NCT04463342
Title: Evaluation of Clinical Performance for Recently Introduced Non Coated Glass Ionomer in Occlusal Caries in Posterior Teeth Compared to Conventional Glass Ionomer With Coating: A Randomized Clinical Trial
Brief Title: Evaluation of Clinical Performance for Recent Non Coated Glass Ionomer in Posterior Teeth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Magdy Eldamanhoury, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU-MMEldamanhoury
Record Dates: First submitted 2020-06-24; First posted 2020-07-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Occlusal Caries
Keywords: Occlusal Caries; Glass Ionomer; Tooth colored Restoration; Non-Coated Glass Ionomer; Universal Glass Ionomer

STUDY DESIGN:
Intervention Model Description: Occlusal Caries in Posterior teeth
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blinded (Participant and Outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Coated Glass Ionomer (Experimental): A faster, easier procedure is great, but you want assurance that reducing chair time doesn't mean compromising on performance. KetacTM Universal AplicapTM Glass Ionomer Restorative saves time by eliminating the need for a coating-yet still delivers the compressive strength and surface hardness that are higher than several competitive glass ionomers which require one.This advancement is the latest in 3M's 30-year history of developing proven and trusted glass ionomers.
  Interventions: Combination Product: Non Coated Glass Ionomer
- Conventional Glass Ionomer with Coat (Active Comparator): A bulk-fill, packable and fast-setting conventional glass ionomer. Because it's less "technique sensitive" than a composite it's ideal for difficult-to-isolate posterior restoration. High compressive strength and marginal integrity make it a glass ionomer of choice for posterior restorations.Ketac Conditioner Dentin Pretreatment is required; Ketac Glaze Light-Cured Varnish applied on the top of the restoration to avoid moisture contamination.
  Interventions: Combination Product: Conventional Glass Ionomer with Coat

INTERVENTIONS:
Combination Product: Non Coated Glass Ionomer — KetacTM Universal AplicapTM Glass Ionomer Restorative saves time by eliminating the need for a coating-yet still delivers the compressive strength and surface hardness that are higher than several competitive glass ionomers which require one.
  Other Names: Ketac Universal Aplicap- Glass Ionomer Restorative
  Arms: Non Coated Glass Ionomer
Combination Product: Conventional Glass Ionomer with Coat — Conventional Glass Ionomer with Coat
  Arms: Conventional Glass Ionomer with Coat

SUMMARY:
In patients with occlusal caries in posterior teeth, does the use of recently introduced non coated glass ionomer provide better clinical performance compared to conventional glass ionomer with surface coating?

-Primary objective: To evaluate clinical performance of different types of restorations (Ketac molar with coating and Ketac Universal Aplicap 3M without coating) in occlusal caries in posterior teeth.

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University; The operator in charge will be Mahmoud Magdy Eldamanhory

Patients will be selected from the outpatient clinic of the department Conservative Dentistry Department, Faculty of Dentistry, Cairo University

* Local anesthesia will be applied to patients complaining about pain or sensitivity to prevent discomfort during restorative procedures.
* Conservative cavity design will be used according to the principals of minimal invasive dentistry.
* All the cavities will be performed by the main author using #57 straight plain carbide fissure bur held in high speed contra-angled hand piece with water cooling system.
* All internal line angles will be slightly rounded.
* Each bur will be discarded after 5 preparations
* If deep caries will be found, it will be removed with large round bur at low speed and a thin layer of calcium hydroxide will be placed on the deep portion of the cavity.
* Isolation will be maintained by using Rubber Dam.
* The dentin and enamel of cavities will be conditioned with 20% polyacrylic acid for 20 seconds (Cavity Conditioner, GC), washed, and briefly dried.
* The restorations will inject into the cavity.
* After the passage of the manufacturer's recommended setting time of 2.5 minutes, the restoration will be trimmed and polished wet using high-speed fine diamonds.

In control group ketac molar with coating:

-After the restoration will briefly dry, Ketac Coat will be applied and photocured for 20 seconds using a photo-curing light.

In study group " Ketac Universal Aplicap 3M without coating":

-The newest addition to glass ionomer family, Ketac Universal Aplicap glass ionomer restorative is a self-cure, one-step placement material designed to help to finish faster. There's no need for conditioning, coating or light-curing steps.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 2 carious class I in same patient.
* The absence of tooth mobility.
* Presence of contact with opposite teeth without any abnormal occlusion stress for the selected teeth.
* Accessible isolation and observable and easily accessible.

Exclusion Criteria:

1. Patients with poor oral hygiene. According to DMF or ADA criteria.
2. The presence of any para functional habit.
3. Abnormal occlusion.
4. Any regurgitation problem.
5. Subjects with compromised medical history.
6. Pulpitis, non-vital or endodontically treated teeth.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Distance penetrated by the Explorer at the tooth restoration interface | during procedure
  The explorer will be drawn across the surface of the restoration toward the tooth
Distance penetrated by the Explorer at the tooth restoration interface | 3 months
  The explorer will be drawn across the surface of the restoration toward the tooth
Distance penetrated by the Explorer at the tooth restoration interface | 6 months
  The explorer will be drawn across the surface of the restoration toward the tooth
Distance penetrated by the Explorer at the tooth restoration interface | 12 months
  The explorer will be drawn across the surface of the restoration toward the tooth
The degree of mismatch from the normal range of tooth shades and translucency | during procedure
  Visual inspection to check the proximity of the shade from the natural tooth
The degree of mismatch from the normal range of tooth shades and translucency | 3 months
  Visual inspection to check the proximity of the shade from the natural tooth
The degree of mismatch from the normal range of tooth shades and translucency | 6 months
  Visual inspection to check the proximity of the shade from the natural tooth
The degree of mismatch from the normal range of tooth shades and translucency | 12 months
  Visual inspection to check the proximity of the shade from the natural tooth
Distance penetrated along the restoration in a pulpal direction | during procedure
  Visual Inspection of the marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure
Distance penetrated along the restoration in a pulpal direction | 3 months
  Visual Inspection of the marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure
Distance penetrated along the restoration in a pulpal direction | 6 months
  Visual Inspection of the marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure
Distance penetrated along the restoration in a pulpal direction | 12 months
  Visual Inspection of the marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | during procedure
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | 3 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | 6 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | 12 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Area of continuous movement of an explorer across the surface of the restoration | during procedure
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Area of continuous movement of an explorer across the surface of the restoration | 3 months
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Area of continuous movement of an explorer across the surface of the restoration | 6 months
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Area of continuous movement of an explorer across the surface of the restoration | 12 months
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Distance seen when the side of the explorer is placed tangentially across the restoration, by which it is not touching two opposing cavosurface line angles at the same time. | during procedure
  Visual inspection and explorer to check the shape and structure of the restoration
Distance seen when the side of the explorer is placed tangentially across the restoration, by which it is not touching two opposing cavosurface line angles at the same time. | 3 months
  Visual inspection and explorer to check the shape and structure of the restoration
Distance seen when the side of the explorer is placed tangentially across the restoration, by which it is not touching two opposing cavosurface line angles at the same time. | 6 months
  Visual inspection and explorer to check the shape and structure of the restoration
Distance seen when the side of the explorer is placed tangentially across the restoration, by which it is not touching two opposing cavosurface line angles at the same time. | 12 months
  Visual inspection and explorer to check the shape and structure of the restoration
Pain due to dentin hypersensitivity (evaporative stimulus) | during procedure
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Pain due to dentin hypersensitivity (evaporative stimulus) | 3 months
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Pain due to dentin hypersensitivity (evaporative stimulus) | 6 months
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Pain due to dentin hypersensitivity (evaporative stimulus) | 12 months
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Eldamanhoury, Master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: expecting to have all the data during January or February 2021
Access Criteria: IPD through contacting the main author Mahmoud.eldamanhory@dentistry.cu.edu.eg.com
URL: http://erepository.cu.edu.eg/index.php/cutheses